CLINICAL TRIAL: NCT00496691
Title: HIV Prevention for Youth With Severe Mental Illness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Dr. Larry K. Brown, Principal Investigator, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01-MH63008-5; R01MH063008 (NIH)
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2015-01

CONDITIONS: HIV Infections
Keywords: HIV prevention; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Parent-child
  Interventions: Behavioral: Family-based HIV prevention program
- 2 (Active Comparator): Adolescent only intervention focusing on condom use skills and assertiveness training around sexual discussions
  Interventions: Behavioral: Family-based HIV prevention program
- 3 (Placebo Comparator): Health promotion intervention including general health promotion topics such as smoking, diet, exercise, etc.
  Interventions: Behavioral: Family-based HIV prevention program

INTERVENTIONS:
Behavioral: Family-based HIV prevention program — comparison between parent-child intervention targeting parent-teen sexual communication, condom use skills, and assertiveness training to an adolescent-only intervention that targets similar constructs minus parent-teen sexual communication and a general health promotion intervention

SUMMARY:
This 4-year competing continuation will extend the follow-up for 750 subjects enrolled in a randomized interventions trial, Project STYLE: "HIV Prevention for Youth with Severe Mental Illness" (R01, MH 63008). Extending the follow-up from one year to 36 months will 1) discern the long-term impact of the Project STYLE interventions and 2) permit complex modeling of the predictors and trajectories of sexual health (delay of sex) and risk (incident STIs). Adolescents, particularly those in mental health treatment, are at risk for HIV because of sexual and substance behaviors. Parent-child communication about sexual topics and parental supervision are associated with delays in the onset of sexual activity and more responsible sexual behavior; thus, the parent project, Project STYLE, is a randomized trial that is evaluating the comparative efficacy of three interventions: a) family-based HIV prevention intervention, b) adolescent-only HIV prevention intervention, and c) general health promotion intervention. This multi-site project (Rhode Island Hospital, Emory University, and the University of Illinois at Chicago) is enrolling an ethnically/racially/geographically diverse group of 750 adolescents in outpatient mental health treatment and their parents. Subjects receive a full day group intervention on the day of randomization, return in two weeks for an individual session, participate in a half day booster session three months later, and are assessed six and 12 months after the intervention. This application offers a unique opportunity to assess this already ascertained sample at three additional points (24,30, and 36 months). This is important because few studies have examined the longer-term predictors of the delay of sex and incident STIs over 36 months using a comprehensive array of family functioning, family monitoring/communication, and trauma history. Additionally, this continuation will provide important data concerning the long-term impact of Project STYLE's theoretically based HIV prevention programs which are designed to maintain safe sexual behaviors. The Family-Based program has increased parent/adolescent sexual communication and reduced adolescent unprotected sex after six months and extended assessment will determine whether these benefits are maintained over time.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent in mental health treatment
* Living with parent/caregiver past 3 months

Exclusion Criteria:

* Adolescent is HIV positive
* Adolescent is pregnant

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 718 (Actual)
Dates: Start 2002-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
condom use; sexual delay | 3 years

SECONDARY OUTCOMES:
parent-adolescent sexual communication | 3 years
condom use attitudes | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Larry K Brown, MD, Principal Investigator — Rhode Island Hospital/ Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Brown LK, Hadley W, Donenberg GR, DiClemente RJ, Lescano C, Lang DM, Crosby R, Barker D, Oster D. Project STYLE: a multisite RCT for HIV prevention among youths in mental health treatment. Psychiatr Serv. 2014 Mar 1;65(3):338-44. doi: 10.1176/appi.ps.201300095. PMID 24382603